CLINICAL TRIAL: NCT03338803
Title: Real World Glycemic Effectiveness of Linagliptin Among Type 2 Diabetes Mellitus Adults by Age and Renal Function
Brief Title: Real World Glycemic Effectiveness of Linagliptin
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218-0182
Record Dates: First submitted 2017-11-08; First posted 2017-11-09 (Actual); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with a written prescription for linagliptin
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — drug
  Other Names: ONDERO, TRAJENTA, TRAYENTA, TRAZENTA, TRADJENTA

SUMMARY:
A non-interventional cohort study using existing data from patients in the Optum Clinical Database which contains electronic health record (EHR) data from providers across the United States to determine whether there is comparable effectiveness of linagliptin on glycemic effectiveness

ELIGIBILITY:
Inclusion Criteria:

* ≥ 1 written prescription for linagliptin (Tradjenta®, Jentadueto®, or Jentadueto XR®)in the EHR (electronic health record) data during the identification period
* ≥ 40 years of age based on the year of the index date
* First active date in the EHR is ≥ 180 days prior to the index date
* ≥ 1 diagnosis code representing Type 2 diabetes (T2DM) in the EHR data during the 180-day pre-index period or on the index date
* ≥ 1 HbA1c value during the 180-day pre-index period or on the index date
* ≥ 1 HbA1c value 60 to 180 days after the index date

Exclusion Criteria:

* ≥ 1 written prescription, medication administration or medication history record for linagliptin or other dipeptidyl peptidase (DPP-4) inhibitor in the EHR data during the 180-day pre-index period
* ≥ 1 written prescription or medication administration for a new antihyperglycemic medication other than linagliptin on the index date New antihyperglycemic medication will be defined as a written prescription or medication administration for any antihyperglycemic medication that was not present in the patient's written prescription, medication administration, or medication history records during the 180-day pre-index period.

Individual antihyperglycemic medications will be distinguished by generic name using the column labelled "Medication Name" in Tables 2 through 13. Combination products containing two generic ingredients will be considered as two distinct antihyperglycemic medications Note: This exclusion criterion is designed to exclude patients from the study sample if they start a new antihyperglycemic medication other than linagliptin on the index date. Patients that start a new antihyperglycemic medication in the follow-up period will not be removed from the study sample to avoid creating a biased sample. Addition of a new antihyperglycemic medication during follow-up will be evaluated through the sensitivity analysis described in Section 9.7.4.4. While we will be capturing additions of new therapies, discontinuation of linagliptin is not able to be accurately measured in electronic record data. The electronic record data capture prescriptions written by a prescriber, but it is not possible to know if patients received and adhered to their medication and there are no structured data fields to identify if and when a medication was discontinued by the patient or the provider

* ≥ 1 diagnosis code or procedure code representing renal transplant, solid organ transplant, or bone marrow transplant in the EHR data during the 180-day pre-index period or on the index date
* ≥ 1 diagnosis code representing malignancy in the EHR data during the 180-day preindex period or on the index date

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A non-interventional cohort study using existing data from patients in the Optum Clinical Database which contains electronic health record (EHR) data from providers across the United States to determine whether there is comparable effectiveness of linagliptin on glycemic effectivenes
Sampling Method: Non-Probability Sample
Enrollment: 11001 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optum, Eden Prairie, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional, retrospective cohort study using existing data from patients in the Optum Clinical Database which contains electronic health record (EHR) data for the period of 01 July 2011 through 31 March 2017.
Pre-assignment Details: Type 2 diabetes mellitus (T2DM) patients with written prescription for initiating Linagliptin (Tradjenta®, Jentadueto®, or Jentadueto XR®) were identified during identification period starting on 01 January 2012 and ending on 30 September 2016. Aim was to describe real world glycemic-lowering effectiveness across range of ages and renal function.
Groups:
- Patients With Written Prescription for Initiating Linagliptin: Patients with a first written prescription for linagliptin were identified during an identification period starting on 01 January 2012 and ending on 30 September 2016.
Period: Overall Study
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
Started | 11001
Completed | 11001
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with a written prescription for linagliptin were identified during an identification period starting on 01 January 2012 and ending on 30 September 2016.
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
Number analyzed (Participants) | 11001
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.30 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5603
  Male | 5398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 927
  Not Hispanic or Latino | 9550
  Unknown or Not Reported | 524
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 241
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1455
  White | 8645
  More than one race | 0
  Unknown or Not Reported | 660
Estimated glomerular filtration rate (eGFR) [Number; unit: participants] — Number of participants by study specific estimated glomerular filtration rate (eGFR) categories is presented.
  participants
    <30 | 679
    30 to 44 | 1646
    45 to 59 | 1727
    60 to 89 | 3256
    ≥ 90 | 2603
    eGFR not available | 1090
Age categories [Number; unit: participants] — Number of participants by study specific age categories is presented
  participants
    40 to 54 years | 2325
    55 to 64 years | 3332
    65 to 74 years | 3077
    75 years and above | 2267

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c) Across Age Categories
Description: Change in HbA1c among adults with type 2 diabetes mellitus (T2DM) within the 60 to 180 days following initiation of linagliptin across pre-defined age categories (40 to 54 years, 40 to 54 years, 65 to 74 years and 75+ years).
  Change in HbA1c, was calculated for each patient by subtracting the patient's last (most recent) HbA1c value during the pre-index period (including the index date) from the patient's last (most recent) HbA1c value 60 to 180 days after the index date.
Time Frame: Baseline and 60 to 180 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
Number analyzed (Participants) | 11001
Percentage (%)
  Overall | -0.51 (1.46)
  Age 40 to 54 years: number analyzed (Participants) | 2325
  Age 40 to 54 years | -0.65 (1.65)
  Age 55 to 64 years: number analyzed (Participants) | 3332
  Age 55 to 64 years | -0.59 (1.54)
  Age 65 to 74 years: number analyzed (Participants) | 3077
  Age 65 to 74 years | -0.43 (1.36)
  Age 75+ years: number analyzed (Participants) | 2267
  Age 75+ years | -0.36 (1.21)

2. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c) Across Renal Function Categories
Description: Change in HbA1c among adults with type 2 diabetes mellitus (T2DM) within the 60 to 180 days following initiation of linagliptin across pre-defined renal function categories.
  Change in HbA1c, was calculated for each patient by subtracting the patient's last (most recent) HbA1c value during the pre-index period (including the index date) from the patient's last (most recent) HbA1c value 60 to 180 days after the index date. Renal function categories were presented based on patients with a pre-index estimated glomerular filtration rate (eGFR) value (eGFR<30, eGFR 30 to 44, eGFR 45 to 59, eGFR 60 to 89, eGFR ≥ 90 milliliter/ minute/1.73 meter^2 and eGFR not available).
Time Frame: Baseline and 60 to 180 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
Number analyzed (Participants) | 11001
Percentage (%)
  Overall | -0.51 (1.46)
  eGFR<30: number analyzed (Participants) | 679
  eGFR<30 | -0.22 (1.46)
  eGFR 30 to 44: number analyzed (Participants) | 1646
  eGFR 30 to 44 | -0.33 (1.34)
  eGFR 45 to 59: number analyzed (Participants) | 1727
  eGFR 45 to 59 | -0.47 (1.42)
  eGFR 60 to 89: number analyzed (Participants) | 3256
  eGFR 60 to 89 | -0.55 (1.44)
  eGFR ≥ 90: number analyzed (Participants) | 2603
  eGFR ≥ 90 | -0.70 (1.58)
  eGFR not available: number analyzed (Participants) | 1090
  eGFR not available | -0.45 (1.40)

3. Secondary Outcome: Percentage of Adults With T2DM Who Achieve HbA1c < 7.0% Across the Pre-defined Age Categories
Description: Percentage of adults with T2DM who achieve HbA1c < 7.0% within the 60 to 180 days following initiation of linagliptin across pre-defined age categories (40 to 54 years, 40 to 54 years, 65 to 74 years and 75+ years).
Time Frame: 60 to 180 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
Number analyzed (Participants) | 11001
Percentage of patients (%)
  Overall | 35.72
  Age 40 to 54 years: number analyzed (Participants) | 2325
  Age 40 to 54 years | 30.28
  Age 55 to 64 years: number analyzed (Participants) | 3332
  Age 55 to 64 years | 35.59
  Age 65 to 74 years: number analyzed (Participants) | 3077
  Age 65 to 74 years | 37.89
  Age 75+ years: number analyzed (Participants) | 2267
  Age 75+ years | 38.55

4. Secondary Outcome: Percentage of Adults With T2DM Who Achieve HbA1c < 7.0% Across Renal Function Categories
Description: Percentage of adults with T2DM who achieve HbA1c < 7.0% within the 60 to 180 days following initiation of linagliptin across pre-defined renal function categories. Renal function categories were presented based on patients with a pre-index estimated glomerular filtration rate (eGFR) value (eGFR<30, eGFR 30 to 44, eGFR 45 to 59, eGFR 60 to 89, eGFR ≥ 90 milliliter/ minute /1.73 meter^2 and eGFR not available).
Time Frame: 60 to 180 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
Number analyzed (Participants) | 11001
Percentage of patients (%)
  Overall | 35.72
  eGFR<30: number analyzed (Participants) | 679
  eGFR<30 | 46.69
  eGFR 30 to 44: number analyzed (Participants) | 1646
  eGFR 30 to 44 | 38.88
  eGFR 45 to 59: number analyzed (Participants) | 1727
  eGFR 45 to 59 | 40.19
  eGFR 60 to 89: number analyzed (Participants) | 3256
  eGFR 60 to 89 | 35.75
  eGFR ≥ 90: number analyzed (Participants) | 2603
  eGFR ≥ 90 | 30.12
  eGFR not available: number analyzed (Participants) | 1090
  eGFR not available | 30.37

ADVERSE EVENTS:
Time Frame: Individual safety reporting is not applicable for this study
Description: This is a retrospective observational study using secondary data, in which all patient data will be collected and analyzed in aggregate. Individual patient safety related information will not be captured during this study. Thus, individual safety reporting is not applicable for this study.
Arm/Group | Patients With Written Prescription for Initiating Linagliptin
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03338803/Prot_SAP_000.pdf